CLINICAL TRIAL: NCT03112239
Title: Chronic Effects Using Light-Emitting Diode Therapy (LEDT) During a Resistance Exercise Protocol for Moderate to Severe Asthmatic Patients: a Randomized Controlled Clinical Trial.
Brief Title: Chronic Effects Using Light-Emitting Diode Therapy (LEDT) During a Resistance Exercise Protocol for Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fabiano Politti (Unknown); LUCIANA MARIA MALOSA SAMPAIO (Unknown)
Responsible Party: Principal Investigator, Ivan Peres Costa, Physitherapist, Master and PhD student, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERAMG-LED-PL-01
Record Dates: First submitted 2016-12-03; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Resistance Training
Keywords: Asthma; Photobiomodulation; Resistance Training
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- photobiomodulation by active LEDT (Active Comparator): The subjects will be initially pre-evaluated by performing pulmonary function tests, peripheral muscle strength tests, functional capacity tests, physical activity questionnaires and clinical control of asthma, and cardiopulmonary exercise test. After the evaluation, patients will be randomized into two resistance training groups, one of them being associated to the intervention with active photobiomodulation by LEDT to increase peripheral muscle function post resistance training.
  Interventions: Device: Light-Emitting Diode Therapy (LEDT)
- photobiomodulation by Placebo LEDT (Placebo Comparator): The subjects will be initially pre-evaluated by performing pulmonary function tests, peripheral muscle strength tests, functional capacity tests, physical activity questionnaires and clinical control of asthma, and cardiopulmonary exercise test. After the evaluation, patients will be randomized into two resistance training groups, one of them being associated to the intervention with placebo LEDT photobiomodulation to increase peripheral muscle function post resistance training.
  Interventions: Device: Light-Emitting Diode Therapy (LEDT)

INTERVENTIONS:
Device: Light-Emitting Diode Therapy (LEDT) — Light-emitting diode, has effects similar to the photobiomodulation by low-level laser intensity.
  Other Names: photobiomodulation by LEDT

SUMMARY:
The objective of this study is to evaluate the effects of LED phototherapy associated with a resistance training protocol on the peripheral muscle function of moderate to severe asthmatic patients ..

DETAILED DESCRIPTION:
This research project will be prospective, analytical and of the randomized controlled clinical trial type, with blind evaluator. The sample type will be consecutive from Santa Casa de Misericórdia de São Paulo. We will study 30 adults of both sexes with moderate to severe asthma between the ages of 20 and 70, based on the sample calculation of the outcomes of this study.

Adult individuals 20 years of age or older with a diagnosis of moderate to severe asthma of both sexes, attended at the Ambulatory of Difficult Asthma Control of Santa Casa de Misericórdia de São Paulo.

Exclusion terms include subjects diagnosed as having heart disease associated with pulmonary disease, musculoskeletal pathology that may interfere with assessment or exercise, pulmonary hypertension, calcium absorption deficiency, BMI ≥ 30 or difficulty learning.

The subjects will initially be pre-evaluated by performing pulmonary function tests, peripheral muscle strength (1-RM), functional capacity tests, physical activity questionnaires and clinical control of asthma and cardiopulmonary exercise test. After the evaluation, patients will be randomized into two resistance training groups, one of them associated with active LED phototherapy and another LED phototherapy placebo.

The resistance exercise protocol will be performed on the muscles: Pectoral, Large Dorsal, Brachial Biceps, Brachial Triceps, Quadriceps and Tibial Ischia. The intensity will be from 40 to 70% obtained in the 1-RM test with two to three sets of ten repetitions.

The load increase will be performed weekly (5%) according to patient tolerance. After 12 weeks all subjects were reevaluated and the last reevaluation occurred at the end of the training program. Patients will only effectively begin participating in this study after explaining the terms of the survey and by accepting written consent from the ICF.

The mean (in kg) of the resistance training protocol for lower limbs in knee extension of group 1 was 33 ± 13 kg and the mean of group 2 was 46 ± 11 kg. The sample calculation was based on the load of the quadriceps muscle, α = 0.05 and β = 95%, determining a minimum of fourteen individuals for each group. An additional 10% was added to compensate for possible losses during the protocol. Thus a minimum of fifteen individuals will be required for the study.

Linear regression models will be used to evaluate the effect of the LED on the results (absolute change and percentage) and a sensitivity analysis with the values of the results in the revaluation, adjusted by the initial value of each result. The possible correlations between the variables can be evaluated using Pearson's correlation. The level of significance adopted will be p <0.5. The analyzes were performed with SPSS 20 software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a medical outpatient setting less than six months; With a stable clinical picture during three months, ie without exacerbations and with optimized drug therapy.

Signed an informed consent form (TCLE) accepting participation in the research.

Exclusion Criteria:

* Diagnosis of heart disease associated with lung disease, musculoskeletal disease that may interfere with assessment or exercise, pulmonary hypertension, calcium absorption deficiency, BMI ≥ 30, or difficulty learning.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pectoral Muscular Strength by 1RM. | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the pectoral muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).
Major Dorsal Muscular Strength by 1RM | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the major dorsal muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).
Femoral Quadriceps Muscular Strength by 1RM | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the femoral quadriceps muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).
Brachial Triceps Muscular Strength by 1RM | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the brachial triceps muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).
Brachial Biceps Muscular Strength by 1RM | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the brachial biceps muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).
Tibial Ischia Muscular Strength by 1RM | Change from Baseline Peripheral muscular Strength up to 24 weeks.
  Muscle strength will be assessed in the tibial ischia muscle group, using the maximal repetition (1RM) test to quantify the resistance training load (between 60 and 80%).

SECONDARY OUTCOMES:
Functional Capacity by Cardiopulmonary exercise test. | Change from baseline measured by cardiopulmonary exercise test up to 24 weeks.
  The cardiopulmonary test will be performed in an electricomagnetic braking cycle ergometer connected to a system composed of gas analysis module attached to a module flow/wave analyzer and a microcomputer BreezeCardiO2 System. (medical Graphics Corporation - MGC, St. Paul, Mo, USA).
Functional Capacity by Incremental Shuytle Walk Test. | Change from baseline measured by Incremental Shuttle Walk Test distance up to 24 weeks.
  The incremental shuttle walk test was performed based on the original test description. The patient walk from side to side in a space of 10 meters identified by two cones inserted 0.5 from each end to avoid such sudden changes in speed. The participant was instructed to walk from cone to cone in one. A single point that the participant must keep pace and a triple beep indicates the beginning of a new level, the height at which the participant has increased the pace. The test comprised 12 levels, each lasting one minute. The speed of the first level was 1.8 Km/h, with an increase of 0.17 m/s every minute until reaching a top speed of 8.53 Km/h. The test was stopped when the participant was unable to reach the cone before the next beep.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana MM Sampaio, PhD, Study Director — University of Nove de Julho
Locations (1):
- Ivan Peres Costa, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers since there is no third party interest in the data collected.

REFERENCES:
- [Background] Miranda EF, Leal-Junior EC, Marchetti PH, Dal Corso S. Acute effects of light emitting diodes therapy (LEDT) in muscle function during isometric exercise in patients with chronic obstructive pulmonary disease: preliminary results of a randomized controlled trial. Lasers Med Sci. 2014 Jan;29(1):359-65. doi: 10.1007/s10103-013-1359-5. Epub 2013 Jun 7. PMID 23743817
- [Result] Dourado VZ, Tanni SE, Antunes LC, Paiva SA, Campana AO, Renno AC, Godoy I. Effect of three exercise programs on patients with chronic obstructive pulmonary disease. Braz J Med Biol Res. 2009 Mar;42(3):263-71. doi: 10.1590/s0100-879x2009000300007. PMID 19287905